CLINICAL TRIAL: NCT07171216
Title: The Effect of REgulation of PArathyroId hoRmone in Patients With Chronic Kidney Disease to Investigate the Change in Bone Mineral Density (Biskjoldbruskkirtelhormon og knogletæthed Hos Patienter Med Kronisk Nyresygdom)
Brief Title: The Effect of REgulation of PArathyroId hoRmone in Patients With Chronic Kidney Disease to Investigate the Change in Bone Mineral Density
Acronym: REPAIR-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Freja Stæhr Hassager, Medical doctor, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-25038403
Record Dates: First submitted 2025-08-29; First posted 2025-09-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease Mineral and Bone Disorder
Keywords: parathyroid hormone; chronic kidney disease; randomized clinical trial; Activated vitamin D
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Intervention in both treatment groups is used to reach a target of PTH (different levels in different groups, no pre-defined treatment)
Who Masked: Investigator
Masking Description: Investigators will be blinded to the primary endpoint (DEXA-scan and the analysis of this)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTH intensive target (Experimental): Intensive parathyroid hormone target (within interval of lower and upper normal limits = 2,0 - 8,5 µmol/L). In the intensive PTH target group, treatment will be initiated as soon as the PTH rise above the upper limit of normal. Participants in this group will receive treatment to lower PTH level (activated vitamin D, phosphate binder, native vitamin D and calcimetics).
  PTH will be measured as intact PTH with Atellica IM PTH assay at Herlev Hospital laboratory (normal range 2,0 - 8,5 µmol/L).
  Interventions: Other: Treat to target
- PTH liberal target (Experimental): Liberal parathyroid hormone target (< 5 x upper normal limit = 42,5 µmol/L). In the liberal PTH target group, treatment will not be initiated until PTH rise above five times the upper limit of normal. This is expected to be a small part of the participants.
  The cut-off for the liberal PTH target (<5 x upper normal limit) was discussed in the national CKD-MBD group. It is chosen to allow the clinician initiate treatment if PTH reaches unusually high levels, no studies have focussed on PTH-targets before, consequently the cut-off is chosen as part of the pragmatic design.
  Interventions: Other: Treat to target

INTERVENTIONS:
Other: Treat to target — Participants will receive treatment from a "toolbox" depending on the situation to reach the PTH target. Available medication is mirroring what is used in the outpatient clinic setting already (native vitamin D, activated vitamin D, phosphate binders, calcimetics).

SUMMARY:
The prevalence of chronic kidney disease (CKD) in the adult population is estimated to 10%. CKD increases risk of bone fractures, cardiovascular disease and death. The main role of parathyroid hormone (PTH) is to regulate mineral metabolism, including the calcium and phosphate homeostasis. PTH increases as the kidney function declines, and at end stage kidney disease almost all patients have disturbances in the mineral metabolism. Decreasing bone mineral density is associated with risk of fracture, both in background population and in patients with CKD.

For decades, treatment with activated vitamin D, phosphate binders, and calcium supplements has been used for patients with chronic kidney disease and elevated parathyroid hormone, but treatment targets have varied greatly over the years, reflecting the lack of randomized clinical trials with clinical important end points.

The purpose of The REPAIR-CKD trial is to determine if treatment of hyperparathyroidism improves the bone mineral density in patients with chronic kidney disease.

During this trial it will also be evaluated if it is feasible to obtain a difference in PTH levels when targeting two different levels of PTH.

Further this trial will explore if a difference in PTH influences on arterial stiffness, muscle mass, muscle function, bone histology and health related quality of life.

DETAILED DESCRIPTION:
The prevalence of chronic kidney disease (CKD) is estimated to afflict 10 % of the adult population, and it is increasing world-wide. CKD is a devastating disease due to the risk of kidney failure and thereby the need for dialysis or transplantation, but also because the presence of CKD increases the risk of bone fracture, cardiovascular disease and mortality.

Parathyroid hormone (PTH) is a peptide hormone produced by the parathyroid glands(5). The main function of PTH is to regulate mineral metabolism, including the calcium and phosphate homeostasis. PTH increases as the kidney function declines, and at end stage kidney disease almost all patients have disturbances in the mineral metabolism. Treatment with activated vitamin D, phosphate binder and calcium supplementation has been used for more than 30 years to suppress hyperparathyroidism and keep calcium and phosphate within the normal range. Later calcimetics has been introduced as a treatment for secondary hyperparathyroidism.

The risk of bone fracture is increased in patients with CKD and the risk increases as the kidney function declines. A bone fracture leads to a direct burden on the individual. In addition, the risk of complications after a bone fracture is higher in the CKD population compared to the general population. A fracture also constitutes a significant cost for the society. The increased risk of fracture in patients with CKD is associated to the presence of hyperparathyroidism.

Bone mineral density (BMD) assessed by dual energy x-ray (DXA) scan is a highly used modality to diagnose osteoporosis and future fracture risk in the general population. Bone mineral density associates with the risk of future fracture in patients with CKD. In patients with CKD there is an association between decreasing eGFR and both low BMD and future fracture risk. It is unknown how elevated PTH associates with BMD and its changes at different stages of CKD, and it is unknown if treatment of hyperparathyroidism influence on BMD and fracture risk in patients with CKD.

The risk of cardiovascular mortality, coronary heart disease, heart failure, stroke and peripheral arterial disease increase as the kidney function declines. Elevated PTH associates with an increased risk of cardiovascular disease. However, hyperparathyroidism is tightly connected to the general disturbances in the mineral metabolism in CKD, i.e. hyperphosphatemia and elevated FGF-23, which associate with an increased risk of cardiovascular disease and mortality. Therefore, it is questioned if PTH is directly involved in the pathogenesis of cardiovascular disease, or if the increased risk of cardiovascular disease could be caused by other factors involved in the mineral metabolism. One way to approach precursors of vascular disease is measuring vascular stiffness with pulse wave velocity which is associated with cardiovascular outcomes in patients with CKD.

The active circulating form of vitamin D is 1,25 dihydroxy vitamin D (calcitriol). The level of calcitriol is regulated by the activity of the 1α hydroxylase enzyme located in the kidney. The 1α hydroxylase enzyme hydroxylate 25-hydroxy vitamin D at the 1-position. As kidney function declines the activity of 1α hydroxylase is reduced and thereby the circulating level of calcitriol is reduced. The reduced level of calcitriol, together with hypocalcaemia and hyperphosphatemia, leads to secondary hyperparathyroidism. Activated vitamin D is given to patients with hyperparathyroidism to try lowering PTH. In a randomized placebo-controlled trial with 36 patients with CKD G3-5 the intervention group were treated with active vitamin D, which resulted in a difference in BMD by +4.2% in the spine compared to controls after 18 months (P< 0.05). No clinical trials have aimed to explore the influence of targeting different levels of PTH and the influence on bone mineral density or bone fracture in patients with CKD.

Two randomized placebo-controlled trials aimed to address effect of 1 year of active vitamin D treatment on the left ventricular mass, a surrogate endpoint for development of heart failure. No difference between the treatment groups was found in any of the trials. Cohort studies in dialysis patients have found increased survival in patients treated with active vitamin D, but the result could be biased having the design in mind. One Japanese randomized controlled trial compared alfacalcidol with placebo in 976 patients on dialysis. Of importance, not all the included participants did have hyperparathyroidism. No difference was found in fatal and non-fatal cardiovascular events, additionally no difference was found in risk of fracture during the study. If this finding would have differed in patients with hyperparathyroidism or in patients with earlier stages of kidney disease and thereby preventable progression of vascular calcification, remains to be determined.

Treatment with active vitamin D, phosphate binders and calcimetics has been used for patients with CKD for decades. Recommendations regarding the appropriate dose and PTH target for different stages of CKD has varied during years and between guidelines, reflecting the lack of randomized clinical trials with clinical important end points.

In patients with CKD G3b-5, it is currently recommended to monitor the PTH every 3-6 month. As more than 50 % of the patients have elevated PTH already at CKD G3b, it is an everyday consideration for the clinician if the patients should be treated to reduce PTH. This is both time- and cost consuming. At present, there is no evidence to advise if secondary hyperparathyroidism should be treated in patients with CKD.

To improve knowledge about when secondary hyperparathyroidism should be treated, investigators want to conduct a randomized clinical trial with one group of patients being treated if PTH is elevated versus a second group of patients not being treated if PTH is elevated.

The investigators hypothesize that suppression of initially elevated PTH will improve BMD, arterial stiffness, muscle mass and muscle strength in patients with CKD.

Subjects will be recruited from the patient population in the outpatient clinic at the Department of Nephrology at Herlev and Gentofte Hospital, Herlev, Denmark.

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years of age at screening
2. CKD G4-5nonD (eGFR < 30 mL/min/1.73m2) based on local laboratory assessment of serum creatinine and eGFR estimated by the CKD-EPI formula)
3. Plasma PTH > upper normal limit of local laboratory reference range (> 8,5µmol/L) and/or treated with active vitamin D (Alphacalcidol) or calcimetics (Cinacalcet) initially
4. Written informed consent

Exclusion Criteria:

1. Patients who have received a kidney transplant
2. Patients receiving treatment with specific anti-osteoporosis medication (denosumab/bisphosphonates) (because of the profound effect on calcium/phosphate fluxes and BMD)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in percent change in bone mineral density (BMD) between the treatment groups. | From baseline to final follow-up at 18 months
  Measured with DEXA-scan

SECONDARY OUTCOMES:
Difference in follow-up BMD between treatment groups | From baseline to final follow-up at 18 months
  Measured with DEXA-scan
Difference in follow-up arterial stiffness between the treatment groups | From baseline to final follow-up at 18 months
  Measured as pulse wave velocity by applanation tonometry with Sphygmocor
Difference in follow-up muscle mass between the treatment groups | From baseline to final follow-up at 18 months
  Measured as appendicular lean body mass (DEXA-scan) as an approximation of muscle mass
Difference in follow-up hand grip strenght between the treatment groups | From baseline to final follow-up at 18 months
  Muscle function will be assessed by different measures including hand grip strenght.
Difference in follow-up 10 meter walk test between the treatment groups | From baseline to final follow-up at 18 months
  Muscle function will be assessed by different measures including 10 meter walk test.
Difference in follow-up sit-to-stand test between the treatment groups | From baseline to final follow-up at 18 months
  Muscle function will be assessed by different measures including sit-to-stand test.
Differences in bone histology between the treatment groups | Labelling at baseline and repeated labelling and biopsy at 18 months
  Tetracycline labelled bone biopsy is performed by a trained physician experienced in performing bone biopsies from the iliac crest after a standardised procedure. At randomisation, we will start with a single labelling of the bone with tetracycline, for us to be able to tell how the bone was at the time of randomisation. Before the biopsy procedure the bone is again labelled with tetracycline
Differences in follow-up health-related quality of life between the treatment groups | From baseline to final follow-up at 18 months
  Health related quality of life will be evaluated through questionnaire "Kidney Disease and Quality of Life" (KDQOL-SF1.3, Danish version).
Differences in number of spinal fractures between the treatment groups | From baseline to final follow-up at 18 months
  Evaluated with DEXA-scan

OTHER OUTCOMES:
The feasibility to obtain a differential PTH level of at least 0.5 times the upper limit of normal between the two groups will be determined | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, Medical doctor, professor, Study Director — Department of Nephrology, Herlev Hospital
Locations (1):
- Department of Nephrology, outpatient clinic, Herlev Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD as the trial will be conducted according to local legislation (Databeskyttelsesloven, Databeskyttelsesforordningen and Sundhedsloven), which does not allow sharing data.

REFERENCES:
- [Background] Rao SD, Matkovic V, Duncan H. Transiliac bone biopsy. Complications and diagnostic value. Henry Ford Hosp Med J. 1980;28(2-3):112-5. No abstract available. PMID 7287505
- [Background] Blake GM, Naeem M, Boutros M. Comparison of effective dose to children and adults from dual X-ray absorptiometry examinations. Bone. 2006 Jun;38(6):935-42. doi: 10.1016/j.bone.2005.11.007. Epub 2005 Dec 22. PMID 16376161
- [Background] Njeh CF, Fuerst T, Hans D, Blake GM, Genant HK. Radiation exposure in bone mineral density assessment. Appl Radiat Isot. 1999 Jan;50(1):215-36. doi: 10.1016/s0969-8043(98)00026-8. PMID 10028639
- [Background] https://www.fda.gov/media/175746/download
- [Background] Frimodt-Moller M, Nielsen AH, Kamper AL, Strandgaard S. Reproducibility of pulse-wave analysis and pulse-wave velocity determination in chronic kidney disease. Nephrol Dial Transplant. 2008 Feb;23(2):594-600. doi: 10.1093/ndt/gfm470. Epub 2007 Nov 7. PMID 17989106
- [Background] Saag KG, Petersen J, Brandi ML, Karaplis AC, Lorentzon M, Thomas T, Maddox J, Fan M, Meisner PD, Grauer A. Romosozumab or Alendronate for Fracture Prevention in Women with Osteoporosis. N Engl J Med. 2017 Oct 12;377(15):1417-1427. doi: 10.1056/NEJMoa1708322. Epub 2017 Sep 11. PMID 28892457
- [Background] Malluche HH, Monier-Faugere MC, Blomquist G, Davenport DL. Two-year cortical and trabecular bone loss in CKD-5D: biochemical and clinical predictors. Osteoporos Int. 2018 Jan;29(1):125-134. doi: 10.1007/s00198-017-4228-4. Epub 2017 Oct 9. PMID 28993865
- [Background] Kang DH, Park CH, Kim HW, Park JT, Han SH, Kim J, Jeong JC, Kim Y, Kim SW, Oh KH, Kang SW, Yoo TH. Kidney function and bone mineral density in chronic kidney disease patients. Clin Kidney J. 2024 Aug 13;17(9):sfae248. doi: 10.1093/ckj/sfae248. eCollection 2024 Sep. PMID 40034486
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Work Group. KDIGO clinical practice guideline for the diagnosis, evaluation, prevention, and treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl. 2009 Aug;(113):S1-130. doi: 10.1038/ki.2009.188. PMID 19644521
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420
- [Background] J-DAVID Investigators; Shoji T, Inaba M, Fukagawa M, Ando R, Emoto M, Fujii H, Fujimori A, Fukui M, Hase H, Hashimoto T, Hirakata H, Honda H, Hosoya T, Ikari Y, Inaguma D, Inoue T, Isaka Y, Iseki K, Ishimura E, Itami N, Ito C, Kakuta T, Kawai T, Kawanishi H, Kobayashi S, Kumagai J, Maekawa K, Masakane I, Minakuchi J, Mitsuiki K, Mizuguchi T, Morimoto S, Murohara T, Nakatani T, Negi S, Nishi S, Nishikawa M, Ogawa T, Ohta K, Ohtake T, Okamura M, Okuno S, Shigematsu T, Sugimoto T, Suzuki M, Tahara H, Takemoto Y, Tanaka K, Tominaga Y, Tsubakihara Y, Tsujimoto Y, Tsuruya K, Ueda S, Watanabe Y, Yamagata K, Yamakawa T, Yano S, Yokoyama K, Yorioka N, Yoshiyama M, Nishizawa Y. Effect of Oral Alfacalcidol on Clinical Outcomes in Patients Without Secondary Hyperparathyroidism Receiving Maintenance Hemodialysis: The J-DAVID Randomized Clinical Trial. JAMA. 2018 Dec 11;320(22):2325-2334. doi: 10.1001/jama.2018.17749. PMID 30535217
- [Background] Teng M, Wolf M, Ofsthun MN, Lazarus JM, Hernan MA, Camargo CA Jr, Thadhani R. Activated injectable vitamin D and hemodialysis survival: a historical cohort study. J Am Soc Nephrol. 2005 Apr;16(4):1115-25. doi: 10.1681/ASN.2004070573. Epub 2005 Feb 23. PMID 15728786
- [Background] Thadhani R, Appelbaum E, Pritchett Y, Chang Y, Wenger J, Tamez H, Bhan I, Agarwal R, Zoccali C, Wanner C, Lloyd-Jones D, Cannata J, Thompson BT, Andress D, Zhang W, Packham D, Singh B, Zehnder D, Shah A, Pachika A, Manning WJ, Solomon SD. Vitamin D therapy and cardiac structure and function in patients with chronic kidney disease: the PRIMO randomized controlled trial. JAMA. 2012 Feb 15;307(7):674-84. doi: 10.1001/jama.2012.120. PMID 22337679
- [Background] Wang AY, Fang F, Chan J, Wen YY, Qing S, Chan IH, Lo G, Lai KN, Lo WK, Lam CW, Yu CM. Effect of paricalcitol on left ventricular mass and function in CKD--the OPERA trial. J Am Soc Nephrol. 2014 Jan;25(1):175-86. doi: 10.1681/ASN.2013010103. Epub 2013 Sep 19. PMID 24052631
- [Background] Rix M, Eskildsen P, Olgaard K. Effect of 18 months of treatment with alfacalcidol on bone in patients with mild to moderate chronic renal failure. Nephrol Dial Transplant. 2004 Apr;19(4):870-6. doi: 10.1093/ndt/gfg595. PMID 15031343
- [Background] Mizobuchi M, Ogata H, Koiwa F. Secondary Hyperparathyroidism: Pathogenesis and Latest Treatment. Ther Apher Dial. 2019 Aug;23(4):309-318. doi: 10.1111/1744-9987.12772. Epub 2018 Dec 18. PMID 30411503
- [Background] https://www.kidney.org/sites/default/files/02-10-4899_GB_SHPT-PTH_v8.pdf
- [Background] Juppner H. Phosphate and FGF-23. Kidney Int Suppl. 2011 Apr;79(121):S24-7. doi: 10.1038/ki.2011.27. Epub 2011 Feb 23. PMID 21346724
- [Background] Brown AJ, Dusso A, Slatopolsky E. Vitamin D. Am J Physiol. 1999 Aug;277(2):F157-75. doi: 10.1152/ajprenal.1999.277.2.F157. PMID 10444570
- [Background] Blacher J, Safar ME, Pannier B, Guerin AP, Marchais SJ, London GM. Prognostic significance of arterial stiffness measurements in end-stage renal disease patients. Curr Opin Nephrol Hypertens. 2002 Nov;11(6):629-34. doi: 10.1097/00041552-200211000-00010. PMID 12394609
- [Background] Palmer SC, Hayen A, Macaskill P, Pellegrini F, Craig JC, Elder GJ, Strippoli GF. Serum levels of phosphorus, parathyroid hormone, and calcium and risks of death and cardiovascular disease in individuals with chronic kidney disease: a systematic review and meta-analysis. JAMA. 2011 Mar 16;305(11):1119-27. doi: 10.1001/jama.2011.308. PMID 21406649
- [Background] Gutierrez OM, Mannstadt M, Isakova T, Rauh-Hain JA, Tamez H, Shah A, Smith K, Lee H, Thadhani R, Juppner H, Wolf M. Fibroblast growth factor 23 and mortality among patients undergoing hemodialysis. N Engl J Med. 2008 Aug 7;359(6):584-92. doi: 10.1056/NEJMoa0706130. PMID 18687639
- [Background] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Background] Matsushita K, Coresh J, Sang Y, Chalmers J, Fox C, Guallar E, Jafar T, Jassal SK, Landman GW, Muntner P, Roderick P, Sairenchi T, Schottker B, Shankar A, Shlipak M, Tonelli M, Townend J, van Zuilen A, Yamagishi K, Yamashita K, Gansevoort R, Sarnak M, Warnock DG, Woodward M, Arnlov J; CKD Prognosis Consortium. Estimated glomerular filtration rate and albuminuria for prediction of cardiovascular outcomes: a collaborative meta-analysis of individual participant data. Lancet Diabetes Endocrinol. 2015 Jul;3(7):514-25. doi: 10.1016/S2213-8587(15)00040-6. Epub 2015 May 28. PMID 26028594
- [Background] Matsushita K, Ballew SH, Coresh J, Arima H, Arnlov J, Cirillo M, Ebert N, Hiramoto JS, Kimm H, Shlipak MG, Visseren FLJ, Gansevoort RT, Kovesdy CP, Shalev V, Woodward M, Kronenberg F; Chronic Kidney Disease Prognosis Consortium. Measures of chronic kidney disease and risk of incident peripheral artery disease: a collaborative meta-analysis of individual participant data. Lancet Diabetes Endocrinol. 2017 Sep;5(9):718-728. doi: 10.1016/S2213-8587(17)30183-3. Epub 2017 Jul 14. PMID 28716631
- [Background] Chen H, Lips P, Vervloet MG, van Schoor NM, de Jongh RT. Association of renal function with bone mineral density and fracture risk in the Longitudinal Aging Study Amsterdam. Osteoporos Int. 2018 Sep;29(9):2129-2138. doi: 10.1007/s00198-018-4592-8. Epub 2018 Jun 15. PMID 29947873
- [Background] Yenchek RH, Ix JH, Shlipak MG, Bauer DC, Rianon NJ, Kritchevsky SB, Harris TB, Newman AB, Cauley JA, Fried LF; Health, Aging, and Body Composition Study. Bone mineral density and fracture risk in older individuals with CKD. Clin J Am Soc Nephrol. 2012 Jul;7(7):1130-6. doi: 10.2215/CJN.12871211. Epub 2012 Apr 19. PMID 22516286
- [Background] Evenepoel P, Cunningham J, Ferrari S, Haarhaus M, Javaid MK, Lafage-Proust MH, Prieto-Alhambra D, Torres PU, Cannata-Andia J; European Renal Osteodystrophy (EUROD) workgroup, an initiative of the CKD-MBD working group of the ERA-EDTA, and the committee of Scientific Advisors and National Societies of the IOF. European Consensus Statement on the diagnosis and management of osteoporosis in chronic kidney disease stages G4-G5D. Nephrol Dial Transplant. 2021 Jan 1;36(1):42-59. doi: 10.1093/ndt/gfaa192. PMID 33098421
- [Background] Jain RK, Vokes T. Dual-energy X-ray Absorptiometry. J Clin Densitom. 2017 Jul-Sep;20(3):291-303. doi: 10.1016/j.jocd.2017.06.014. Epub 2017 Jul 14. PMID 28716497
- [Background] Xu Y, Evans M, Soro M, Barany P, Carrero JJ. Secondary hyperparathyroidism and adverse health outcomes in adults with chronic kidney disease. Clin Kidney J. 2021 Jan 20;14(10):2213-2220. doi: 10.1093/ckj/sfab006. eCollection 2021 Oct. PMID 34603697
- [Background] Borgstrom F, Zethraeus N, Johnell O, Lidgren L, Ponzer S, Svensson O, Abdon P, Ornstein E, Lunsjo K, Thorngren KG, Sernbo I, Rehnberg C, Jonsson B. Costs and quality of life associated with osteoporosis-related fractures in Sweden. Osteoporos Int. 2006;17(5):637-50. doi: 10.1007/s00198-005-0015-8. Epub 2005 Nov 9. PMID 16283064
- [Background] Runesson B, Trevisan M, Iseri K, Qureshi AR, Lindholm B, Barany P, Elinder CG, Carrero JJ. Fractures and their sequelae in non-dialysis-dependent chronic kidney disease: the Stockholm CREAtinine Measurement project. Nephrol Dial Transplant. 2020 Nov 1;35(11):1908-1915. doi: 10.1093/ndt/gfz142. PMID 31361316
- [Background] Hansen D, Olesen JB, Gislason GH, Abrahamsen B, Hommel K. Risk of fracture in adults on renal replacement therapy: a Danish national cohort study. Nephrol Dial Transplant. 2016 Oct;31(10):1654-62. doi: 10.1093/ndt/gfw073. Epub 2016 Apr 19. PMID 27190324
- [Background] Naylor KL, McArthur E, Leslie WD, Fraser LA, Jamal SA, Cadarette SM, Pouget JG, Lok CE, Hodsman AB, Adachi JD, Garg AX. The three-year incidence of fracture in chronic kidney disease. Kidney Int. 2014 Oct;86(4):810-8. doi: 10.1038/ki.2013.547. Epub 2014 Jan 15. PMID 24429401
- [Background] Komaba H, Nakanishi S, Fujimori A, Tanaka M, Shin J, Shibuya K, Nishioka M, Hasegawa H, Kurosawa T, Fukagawa M. Cinacalcet effectively reduces parathyroid hormone secretion and gland volume regardless of pretreatment gland size in patients with secondary hyperparathyroidism. Clin J Am Soc Nephrol. 2010 Dec;5(12):2305-14. doi: 10.2215/CJN.02110310. Epub 2010 Aug 26. PMID 20798251
- [Background] Hansen D. A randomised clinical study of alfacalcidol and paricalcitol. Dan Med J. 2012 Feb;59(2):B4400. PMID 22293059
- [Background] Levin A, Bakris GL, Molitch M, Smulders M, Tian J, Williams LA, Andress DL. Prevalence of abnormal serum vitamin D, PTH, calcium, and phosphorus in patients with chronic kidney disease: results of the study to evaluate early kidney disease. Kidney Int. 2007 Jan;71(1):31-8. doi: 10.1038/sj.ki.5002009. Epub 2006 Nov 8. PMID 17091124
- [Background] Goodman WG, Quarles LD. Development and progression of secondary hyperparathyroidism in chronic kidney disease: lessons from molecular genetics. Kidney Int. 2008 Aug;74(3):276-88. doi: 10.1038/sj.ki.5002287. Epub 2007 Jun 13. PMID 17568787
- [Background] Goltzman D. Physiology of Parathyroid Hormone. Endocrinol Metab Clin North Am. 2018 Dec;47(4):743-758. doi: 10.1016/j.ecl.2018.07.003. Epub 2018 Oct 11. PMID 30390810
- [Background] Moe SM, Drueke T, Lameire N, Eknoyan G. Chronic kidney disease-mineral-bone disorder: a new paradigm. Adv Chronic Kidney Dis. 2007 Jan;14(1):3-12. doi: 10.1053/j.ackd.2006.10.005. PMID 17200038
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Xie Y, Bowe B, Mokdad AH, Xian H, Yan Y, Li T, Maddukuri G, Tsai CY, Floyd T, Al-Aly Z. Analysis of the Global Burden of Disease study highlights the global, regional, and national trends of chronic kidney disease epidemiology from 1990 to 2016. Kidney Int. 2018 Sep;94(3):567-581. doi: 10.1016/j.kint.2018.04.011. Epub 2018 Aug 3. PMID 30078514

DOCUMENTS (1):
  • Study Protocol (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT07171216/Prot_000.pdf